CLINICAL TRIAL: NCT03326778
Title: Register Zur Erhebung Von Langzeitergebnissen Nach Chirurgischem Aortenklappen Ersatz Mit Einer "Rapid Deployment" Aortenklappenprothese (Edwards Intuity) in Kombination Mit Einer Bypassoperation (CABG)
Brief Title: Registry to Gather Long-time Results After Surgical Aortic Valve Replacement With a "Rapid Deployment Aortic Valve Prothesis (Edwards Intuity) Combined With Bypss Surgery (CABG)
Acronym: INCA
Status: Completed | Type: Observational
Sponsor: Campus Bad Neustadt (Other)
Collaborators: Edwards Lifesciences (Industry); Software for Trials Europe GmbH (Unknown); Institut für Pharmakologie und Präventive Medizin (Network)
Responsible Party: Sponsor
Other Study IDs: INCA
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Aortic Valve Stenosis; Coronary Artery Disease
Keywords: Aortic Valve Stenosis; Rapid deployment Valve; CABG; Edwards Intuity Elite
MeSH Terms: conditions — Aortic Valve Stenosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- AVR + CABG: Patient receiving AVR combined with CABG
  Interventions: Procedure: AVR and CABG

INTERVENTIONS:
Procedure: AVR and CABG — Combined AVR with CABG

SUMMARY:
This is a prospctive, unrandomized multicentric registry which will enrol patients with an indication for aortc valve replacement combined with myocardial reperfusion (CABG). The registry will collect patient specific baseline data and established risk scores (Logistic Euroscore I & II, STS-Score, KBA Score) to enable us to make an estimate about the perioperative risks.

DETAILED DESCRIPTION:
Aortic replacement combined with coronary bypass surgery has an impact on the risk profile for the direct postoperative course and also on the long-time survival perspective.

The advantage of rapid deployment aortic valve prostheses, like the Edward Intuity Elite Valve that is used in this registry, is the greater ease of implantation, because only a few sutures are necessary to secure the device compared to a conventional prosthesis, where more then ten sutures are needed. In procedures where the aortic valve replacement (AVR) is combined with a coronary artery bypass graft (CABG), the use of a rapid deployment valve can shorten the duration of cardiac ischemia and the overall intervention duration, which possibly has an influence on clinical results.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* patients with aortic valve stenosis and coronary heart disease with indication for AVR and CABG
* patients in who the Edwards Intuity Elite valve is to be implanted
* patients who are planned to receive at least one coronary bypass
* patients who have signed an informed consent form

Exclusion Criteria:

* Exclusion Criteria:
* emergency surgery
* re-operation (i.e. any previous opening of pericardium)
* additional heart diseases requiring heart surgery (e. g. subvalvular myectomy and ablation, but not atrial auricle closure or resection)
* legal incapacity or other circumstances that impair the patient's ability to understand the nature, meaning or extent of the trial
* patients wanting a mechanical prosthesis
* patients with contraindications for the Edwards Intuity Elite Valve
* acute endocarditis or other systemic infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for AVR combined with CABG who will receive an Edwards Intuity Elite rapid deployment aortic valve prosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2017-11-26 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
all-cause mortality | 30 Days
  death from any reason

CONTACTS AND LOCATIONS:
Overall Officials: Anno Diegeler, Prof., Principal Investigator — Campus Bad Neustadt
Locations (1):
- Campus Bad Neustadt, Bad Neustadt an der Saale, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided